CLINICAL TRIAL: NCT07272941
Title: Multisite Randomized Clinical Trial: Mindfulness-Based Intervention for Mild Traumatic Brain Injury (MBI-4-mTBI)
Brief Title: Mindfulness-Based Intervention for Pediatric Mild Traumatic Brain Injury
Acronym: MBI-4-mTBI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: The Hospital for Sick Children (Other); Montreal Children's Hospital of the MUHC (Other); University of Ottawa (Other); British Columbia Children's Hospital (Other); Stollery Children's Hospital (Other)
Responsible Party: Principal Investigator, Andree-Anne Ledoux, Scientist, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 516950; 516950 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Concussions; Mild Traumatic Brain Injury, Concussion; Concussion Mild
Keywords: mild traumatic brain injury; mtbi; concussion; intervention; meditation; quality of life; treatment; Persistent post-concussive symptoms; mindfulness
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Pragmatic-blind randomized clinical trial with two two groups who will be studied: (1) experimental group: usual care plus early introduction of the app-based MBI; and (2) a delayed-start (crossover) control group: usual care plus early introduction sham application, including the cognitive math game called 2048, with option to receive experimental app-based MBI after 4 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Pragmatic-blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Intervention + Usual Care (Experimental): Experimental group: MBI training will consist of a 4-week custom-made program that includes setting intentions and check-in with mood, audio-recorded lectures, guided meditations such as body scans, and writing events journal. Each standardized course will be unlocked as the participant progresses through the program. Users will be encouraged to participate in the app-based activities for a total of 10-15 minutes every day, with a minimum of 4 days a week, over a period of 4 weeks (with the option to continue for 8 weeks).
  Interventions: Behavioral: Mindfulness Based Intervention (MBI)
- Cognitive Sham + Usual care (Sham Comparator): Usual care recommends that patients refrain from physical and cognitive activities for 24-48 hours after concussion. After the initial rest period, it is recommended to introduce low to moderate levels of physical and cognitive activity at a level that does not result in recurrence or exacerbation of symptoms. Patients must refrain from any activities that increase the risk of re-injury (body contact or risk falls) until fully asymptomatic and cleared by their primary care or other medical provider. This arm is considered as active participant with the sham app (cognitive math game called "2048") delivered via the same app as the MBI, but without the mindfulness content. Participants will be encouraged to engage in the app-based activities for at least 10 minutes daily, with a minimum of 4 days per week, over a period of 4 weeks. Participants will also be asked questions about their stress, emotions, and symptoms.
  Interventions: Behavioral: Cognitive Sham

INTERVENTIONS:
Behavioral: Mindfulness Based Intervention (MBI) — Using the Dawn MBI-based app, targeted MBI training will consist of a 4-to-8-week custom-made program that includes audio-recorded lectures, guided meditations such as walking meditations and body scans, setting intentions and check-in with mood, and writing events journal. Each standardized course is unlocked as the participant progresses through the MBI program. Participants will be encouraged to engage in the app-based activities for at least 10 minutes every day, with a minimum of 4 days per week, over a period of 4 weeks (with option to continue for 8 weeks).
  Other Names: MBI; Dawn
  Arms: Mindfulness Intervention + Usual Care
Behavioral: Cognitive Sham — Usual care recommends that the patient refrain from physical and cognitive activities for 24-48 hours after injury. After the rest period, it is recommended that low to moderate levels of physical and cognitive activity be gradually started 24-48 hours after injury. The activities should be performed at a level that does not result in recurrence or exacerbation of symptoms. Children must refrain from any activities that increase the risk of re-injury (drills with body contact or that risk falls) until fully asymptomatic and cleared by their primary care or other medical provider. The sham journey will consist of playing an open-source cognitive math game (called "2048") delivered through the same app as MBI, but without the mindfulness content. Participants will be encouraged to utilize the app for at least 10 minutes every day, with a minimum of 4 days a week, over a period of 4 weeks.
  Other Names: Usual Care
  Arms: Cognitive Sham + Usual care

SUMMARY:
Formal MBIs, such as Mindfulness-Based Stress Reduction (MBSR), have been shown to increase resiliency and teach affect regulation. However, these formal interventions may not be suitable for acutely concussed youth as they are costly, not easily accessible (trained therapists are needed), and require commitment from parents and children for in-person weekly meetings and at-home practice of learned skills for 8 to 16 weeks. Further, MBSR programs may not be readily accessible immediately after a concussion. With the increasing use of mobile phones and tablets in youth, mobile health offers a powerful platform for mental health interventions. Advantages of app-based interventions include constant availability, greater access, tailored content, lower cost, immediate delivery, and increased service capacity and efficiency. Therefore, the anticipated benefit is to show the efficacy of a pragmatic and low-cost intervention and reduce barriers to care through a novel, innovative and accessible MBI treatment program. This will have both a benefit to public health and expand our understanding of the impact of MBIs on pediatric recovery.

DETAILED DESCRIPTION:
The proposed study has two groups: (1) experimental group: usual care plus early introduction of the app-based MBI; and (2) control group: usual care plus early introduction sham application, including the cognitive math game called 2048. Usual care in both groups refers to the recommended return to physical and cognitive activity 24-48 hours post-injury. To maintain valid results, participants will be "blinded" to their intervention. (i.e., during the informed consent process, the study will be referred to as the App-based Intervention study with the purpose of evaluating two app-based interventions). Although only one group will receive the MBI intervention, both groups will be receiving usual care instructions, which involves the early return to cognitive and physical activities. Therefore, both groups will be receiving a beneficial intervention with the experimental group receiving the additional MBI that is being assessed. For both groups, Treatment Coaches will be assigned to each participant. Coaches will maintain regular communication with patients. Their role will be to encourage and assist participants throughout the study duration through a standardized question-and-answer protocol. Additionally, to increase adherence to the intervention, participants will complete a motivational interview at 2 weeks. After 4 weeks, all participants will be offered the MBI program for an extra period of 4 weeks. The control group will have the possibility at that time to crossover and start the intervention if desired.

ELIGIBILITY:
Inclusion Criteria:

* Participants presenting to five PERC EDs after sustaining a direct or indirect head injury
* Aged 12 through 17.99 years
* Diagnosed with a definite or suspected concussion, defined by the American College of Rehabilitation Medicine definition
* Score ≥6 on the 5P rule
* Suffered the index injury in the previous 48 hours
* Proficient in English or French

Exclusion Criteria:

* Glasgow Coma Scale ≤13
* Abnormality on standard neuroimaging studies, including positive head CT findings (Note: neuroimaging is not required, but may be performed if clinically indicated)
* Neurosurgical operative intervention, intubation or intensive care required
* Multi-system injuries with treatment requiring hospital admission, operating room or procedural sedation in ED (Note: hospital admission for observation or management of ongoing concussion symptoms is not an exclusion criteria)
* Severe neurological developmental delay resulting in communication difficulties
* Intellectual disability/mental retardation, autism spectrum disorder (history of attention deficit hyperactivity disorder, learning disability, or Tourette's syndrome is not an exclusion)
* Intoxication at the time of ED presentation as per clinician judgment
* No clear history of trauma as primary events (e.g., seizure, syncope or migraine)
* Prior psychiatric hospitalization
* Prior diagnosis of severe psychiatric disorder such as schizophrenia (diagnosis of anxiety or depression are not exclusionary)
* Inability to obtain a proper written informed consent/assent (language barrier, absence of parental authority, developmental delay, intoxication, patient too confused to consent, etc.)
* Legal guardian not present (certain forms need be completed by parents/legal guardians)
* No internet or mobile/tablet access.
* Previously enrolled in phase 1 or phase 2 of the feasibility trial or the efficacy trial.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 362 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory™ version 4.0 | Day of enrolment (ED), Week 4, Week 8
  The PedsQL is a reliable and valid measure of quality of life (QoL) in healthy children and adolescents and those with acute and/or chronic health conditions. Parent versions exist for children aged 2 to 18 years (in 4 age groups) and child versions for those aged 5 and over. For this study, only the child's version (ages 8-12 and ages 13-18) will be used. The inventory covers four domains: physical, emotional, social, and school, the sum of which is total QoL. This measure will be used to assess whether early brief MBI can improve total QoL. Higher scores indicate better health related to QoL.

SECONDARY OUTCOMES:
Connor-Davidson Resilience Scale-10 (CD-RISC) | Day 1, Week 4, & Week 8
  A Validated measure offered in both English and French for the adolescent concussion population that assesses the individual's own perception of hardiness or perceived stress. It is a 10-item rating scale, 5-point Likert scale; the scale is summed and provides a total score (0-40) for the level of resilience. A lower score is attributed to lesser levels of resilience.
The 18-item PedsQL™ Multidimensional Fatigue Scale (PedsQL-MFS) | Day 1, Week 4, & Week 8
  Designed to measure fatigue in pediatric patients and comprises the General Fatigue Scale (6 items), Sleep-Rest Fatigue Scale (6 items), and Cognitive Fatigue Scale (6 items). The PedsQL™ Multidimensional Fatigue Scale has demonstrated excellent internal consistency, reliability and validity. For this study, only the child's version (ages 8-12 and ages 13-18) will be used. Higher scores are associated with less fatigue.
Health and Behaviour Inventory (HBI) | Day of enrolment (ED; retrospective (parents) and post-injury (participant)), Week 2, Week 4, & Week 8
  This assessment will be used to measure the degree of symptoms, available in both English and French. The HBI is a 20-item self-report questionnaire, Likert scale (0, 1, 2, or 3 points) yielding separate scores for cognitive and somatic symptom scales for a total score range of 0 to 60. Higher scores indicate a higher degree of symptoms. Participants will complete a post-injury measure, while parents will complete a retrospective (pre-injury) measure at an emergency department presentation. Only participants will complete HBI measures at follow-up.
The General Anxiety Disorder 7-items (GAD-7) | Day of enrolment (ED), Week 4, & Week 8
  The GAD-7 is a validated, reliable and sensitive to treatment-related changes tool that assesses anxiety symptoms in youth. It is a 7-item scale, 3-point Likert scale, providing a sum score (0-21) of the level of GAD. A higher score indicates a worse outcome. It is available for participants in both English and French.
Center for Epidemiologic Studies Short Depression Scale (CES-D-10) | Day of enrollment (ED), Week 4, & Week 8
  The CES-D-10 is a 10-item questionnaire assessing how individuals feel during the past week. This is a short version of the 20-item CES-D tool. Graded on a 4-point Likert scale, with items 5 and 8 scored inversely. The final score is the sum of the graded items with higher scores indicating a worse outcome. The CES-D-10 has good internal consistency (Cronbach's α=0.86) and test-retest reliability (I CC=0.85). It is also available in both English and French.
Child and Adolescent Mindfulness Measure (CAMM) | Day 1, Week 4, & Week 8
  The CAMM is a 10-item validated self-report measure of mindfulness for use with children and adolescents, in both English and French. Responses are scored on a 5-point Likert scale. Lower scores indicate higher tendencies to be mindful in everyday life.
Pediatric Fear Avoidance Behavior After Traumatic Brain Injury (PFAB-TBI) | Week 4 & Week 8
  The Pediatric Fear Avoidance Behavior After Traumatic Brain Injury (PFAB-TBI) is a validated measure used in the pediatric population with concussion to measure the degree of fear avoidance as a negative coping style post-injury. It is comprised of 16-item, 4-point Likert scale asking participants to agree with statements that range from 0 ("strongly disagree") through 3 ("strongly agree"). The total item score is out of 48 with higher scores associated with more negative clinical outcomes.(Cairncross et al., 2021). This measure is offered in both English and French.
Avoidance and Fusion Questionnaire for Youth Short Form (AFQ-Y8) | Day 1, Week 4 & Week 8
  The AFQ-Y8 is the 8-item short-form version of the original 17-item AFQ-Y, a self-report measure examining psychological inflexibility in youth. This validated measure comprises two constructs of psychological inflexibility: cognitive fusion (the belief that inner thoughts are true and allow them to dominate behaviour) and experiential avoidance (avoidance or suppression of unwanted internal experiences). Participants are asked to agree with statements on a 5-point Likert scale with responsed from not true at all (0) to very true (4). Items are summed to produce a final score between 0 and 32, with a higher score indicating greater psychological inflexibility. Measures are available in both English and French.
Perceived Stress Scale (PSS-10) | Day of enrollment (ED), Week 4, & Week 8
  A 10-item self-report questionnaire examining an individual's perception of stress. The items are ranked on a 5-point Likert scale, asking participants to respond from Never (1) to very often (5). Items 4, 5 and 7 are positively worded and reverse-scored, then all items are summed. Higher scores indicate that participants are more likely to appraise events as stressful. Participants also have the option to complete the measure in English or French.
Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA) | Day 1, Week 4, & Week 8
  A validated 10-item questionnaire used in adolescent populations to measure emotion regulation. The measure consists of 2 subcategories: cognitive reappraisal (6 items) and expressive suppression (4 items). . Responses to items include a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Composite scores for cognitive reappraisal range from 6-30 and 4 to 20 for expressive suppression. Scores are typically interpreted separately. Higher reappraisal scores are associated with positive tendencies to reframe situations to regulate emotions, while higher repressive scores are negatively associated with the tendency to inhibit emotions. This measure can be completed in English of French.
Credibility Score (Credibility and Expectancy Questionnaire (CEQ)) | Week 1
  The CEQ is a 6-item questionnaire (9-point Likert scale) assessing credibility and expectancy. The validated questionnaire demonstrates excellent reliability across different populations and is available in both English and French. A higher score indicates more credibility.
Modified version of the Client Satisfaction Questionnaire (CSQ) | Week 4
  This is a validated, reliable, 8-item questionnaire used to measure client satisfaction with a particular program or service. In this case, the questionnaire has been modified to assess participant satisfaction with the app-based intervention. It is available to participants in English or French.

OTHER OUTCOMES:
Self assessments | Daily through study completion, on average 8 weeks.
  Upon entering the app, participants will be asked daily to self-asses their mood and levels of stress. Self-assessed stress is captured via a visual-point scale and self-assessed emotions are captured via participant selecting their emotions. There is also a daily thought journal included within the app. requiring participants to journal their thoughts in the moment daily and write their positive thoughts.
Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTAQ) | Week 1, Week 2, Week 4, Week 8
  The GSLTAQ was developed to classify physical activities/exercises performed into three subgroups: strenuous, moderate, and light. The frequency and type of activity/exercise score performed over the past week are used to calculate the physical activity/exercise total score. A higher score corresponds to a higher level of weekly activity/exercise.
Puberty Questionnaire | Day of enrollment (ED)
  The questionnaire is a 5 question, self-administered rating scale for pubertal development without pictorial representations or interviews. Separate forms are used for boys and girls. For Items 1 through 4 on the girls' version and all items on the boys' version, response options are: not yet start (1 point); barely started (2 points); definitely started (3 points); seems complete (4 points); I don't know. Yes, on the menstruation item for girls is 4 points, while No is 1 point. Points are then averaged for all items to give a Pubertal Developmental Scale. Pubertal Category Scores can also be computed.
Return to school and physical activity questions | Week 1, Week 2, Week 4, Week 8
  Participants will be asked if or when they returned to a full day of school, and if or when they have returned to usual levels of physical activity. These questions will be asked at follow-up each week after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Andrée-Anne Ledoux, PhD, Principal Investigator — Children's Hospital of Eastern Ontario Research Institute
Locations (5):
- Canada (5):
  - Stollery Children's Hospital, Edmonton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital of Sick Children (SickKids), Toronto, Ontario
  - BC Children's Hospital, Vancouver, Ontario
  - Montreal Children's Hospital, Montreal

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the study protocol and statistical analysis plan.
Supporting Information: Study Protocol, SAP
Time Frame: These documents will be shared once the protocol is published
Access Criteria: The protocol will be accessible online and through Trial.gov